CLINICAL TRIAL: NCT05275660
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled Study Investigating the Safety, Tolerability, and Pharmacokinetics of Single Dose Intravenously Administered HFB30132A, a Monoclonal Antibody Against SARS-CoV-2, in Chinese Healthy Adult Subjects
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of HFB30132A Against COVID-19 in Chinese Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HiFiBiO Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCSW-XGAB-Ⅰ01
Record Dates: First submitted 2022-03-10; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Healthy
MeSH Terms: interventions — enuzovimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HFB30132A (Experimental): Participants will receive HFB30132A administered across 2 fixed-dose cohorts via intravenous infusions (to be administered sequentially)
  Interventions: Drug: HFB30132A
- Placebo (Placebo Comparator): Placebo will be administered to participants across three fixed-dose cohorts similar to the active treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HFB30132A — Participants randomized to HFB30132A will be administered dose 1 in cohort 1. Participants in Cohort 2 will receive HFB30132A dose 2.
  Arms: HFB30132A
Other: Placebo — Participants randomized to placebo will receive the same volume of solution as participants on active treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety and tolerability of HFB30132A when it is given by single intravenous infusion in Chinese healthy participants.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, placebo-controlled, dose escalation study in Chinese healthy volunteers.

The study will comprise of:

1. A Screening Period of up to 30 days (Day -30 through Day -1);
2. A Treatment Period during which participants will be resident at the Observation Unit from Day -1, 1 day before Investigational Medicinal Product (IMP) administration (on Day 1) until at least 48 hours (Day 3) after IMP administration. Participants will be discharged on Day 3 after all safety and/or pharmacokinetic (PK) evaluations have been completed, and
3. A Follow up Period lasting 270 days after the IMP dose.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy male or female subject, aged between 18 to 60 years (inclusive). A Body Mass Index (BMI) of between 18 to 30 kilograms per square meter (kg/m^2) inclusive, and a body weight of ≥45 kg for female, ≥50 kg for male.
* Health is defined as no clinically relevant abnormalities identified by Investigator's decision based on a detailed medical history, full physical examination, including blood pressure, heart rate, respiratory rate, and body temperature measurement, electrocardiogram (ECG) and clinical laboratory tests prior to the study drug administration.
* Subject voluntarily has given written informed and is willing and able to comply with all scheduled visits, treatment plan, clinical laboratory tests, lifestyle guidelines, methods of contraception
* Female subjects of childbearing potential must not be planning a pregnancy or be pregnant or lactating. All female subjects must have a negative result for the pregnancy tests performed at screening and admission.
* For female subjects of childbearing potential: must agree to use a reliable method of contraception until study completion and for at least 4 weeks following their final study visit
* Female subject of non-childbearing potential defined as surgically sterile (i.e. documented bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or at least 12 months postmenopausal.
* Male subjects with partners of childbearing potential must have had surgical sterilization (vasectomy) at least 26 weeks prior to screening or use a male barrier method of contraception (i.e. male condom with spermicide) during any sexual intercourse, from Study Day -1 (beginning of confinement) until 3 months after the final Follow-up Visit. Note: complete abstinence from sexual intercourse is acceptable.
* Male subjects must agree to abstain from sperm donation from initial study drug administration through 3 months after the last Follow-up Visit.
* Subject voluntarily agrees to participate in this study and has given written informed consent prior to undergoing any of the screening procedures.

Exclusion Criteria:

* History or symptoms of any clinically significant cardiovascular, hepatic, renal, gastrointestinal, neurological, pulmonary, hematological, autoimmune, psychiatric disease, metabolic disorder.
* History of pulmonary tuberculosis and clinically significant abnormal chest CT results
* History of drug or alcohol abuse within 1 year prior to screening, or positive test for drugs of potential abuse at screening and admission, where alcohol abuse is defined as regular consumption exceeding 7 drinks/ week for women, and 14 drinks/ week for men.
* Use of any medications started within 14 days (or 5 half-lives, whichever is longer) prior to study drug administration including, prescription medications, nutritional supplements, and over-the-counter medications
* Blood donation of approximately 500 mL within 60 days prior to dosing, or donation of more than 200 mL within 30 days, or receipt of any transfused blood products within 60 days prior to the screening visit
* Receipt of treatment or vaccination against SARS-CoV-2 within 90 days prior to dosing, or planning for vaccination against SARS-CoV-2 from screening to 90 days after dosing
* Receipt of influenza vaccination within 4 weeks before screening or planning to receive influenza vaccination from screening to 90 days after dosing
* Symptoms of acute respiratory tract infection within 28 days before dosing
* Febrile illness within 28 days prior to the first dose of study drug, or other signs or symptoms consistent with SARS-CoV-2 infection in the judgement of the Investigator in the 14 days prior to the first dose of study drug.
* Hospitalization for any reason within 60 days prior to the screening visit
* Participation (defined as receipt of dose of investigational agent) in any clinical research study evaluating another investigational drug or therapy within 3 months prior to the screening visit
* History of or positive human immunodeficiency virus (HIV) screen result, or positive blood test for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) or subjects with positive hepatitis C virus (HCV) antibody.
* Subject is confirmed as positive by SARS-CoV-2 RT-PCR or antibody testing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-09 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent serious adverse events (TESAEs) | From Day 1 to up to Day 30 after the single dose administration of HFB30132A
  Number of participants experiencing TESAEs
Number of participants with treatment emergent adverse events of special interest (TEAESI) | From Day 1 to up to Day 30 after the single dose administration of HFB30132A
  Safety and tolerability will be evaluated in terms of number of participants with TEAESI (hypersensitivity / anaphylactic reaction / local tolerability)
Number of participants with treatment-emergent adverse events (TEAE) | From Day 1 to up to Day 30 after the single dose administration of HFB30132A
  Safety and tolerability will be evaluated in terms of number of participants with TEAE
Number of participants with changes in laboratory values, vital signs and ECG parameters | From Day 1 to up to Day 30 after the single dose administration of HFB30132A
  Safety and tolerability will be evaluated in terms of number of participants with changes in laboratory values, vital signs and ECG parameters
Maximum observed serum concentration (Cmax) | From Day 1 to up to Day 30 of the last enrolled subject
Time of maximum serum concentration (Tmax) | From Day 1 to up to Day 30 of the last enrolled subject
Area under the concentration vs. time curve (AUC0-last), AUC0-∞) | From Day 1 to up to Day 30 of the last enrolled subject
Terminal half-life (T1/2) | From Day 1 to up to Day 30 of the last enrolled subject
Systemic clearance (CL) | From Day 1 to up to Day 30 of the last enrolled subject
Apparent volume of distribution (Vd) | From Day 1 to up to Day 30 of the last enrolled subject

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Li S, Hedrich W, Wu X, Li S, Qiu C, Lin K, Bian X, He J, Zhou H, Adrian F, Schweizer L, Zhang J. Population pharmacokinetics and pharmacodynamics of HFB30132A, a monoclonal antibody against SARS-CoV-2, in healthy Chinese and US subjects. Int J Antimicrob Agents. 2025 Mar;65(3):107439. doi: 10.1016/j.ijantimicag.2024.107439. Epub 2025 Jan 9. PMID 39793935
- [Derived] Li S, Wu X, Li N, Cao G, Wang J, Chen Y, Li S, He J, Wu J, Yang H, Lin K, Qiu C, Liu A, Zhou H, Adrian F, Schweizer L, Zhang W, Gu J, Zhang J. Safety, tolerability, pharmacokinetics, and immunogenicity of an anti-SARS-CoV-2 monoclonal antibody HFB30132A after single dose intravenous administration in healthy Chinese subjects: a phase 1, randomized, double-blind, placebo-controlled study. Front Pharmacol. 2023 May 23;14:1117293. doi: 10.3389/fphar.2023.1117293. eCollection 2023. PMID 37332355